CLINICAL TRIAL: NCT02307721
Title: Pharmacokinetics and Pharmacodynamics of a New Formulation of Nasal Naloxone for Prehospital Use
Acronym: OPI-14-001
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Norwegian University of Science and Technology (Other)
Collaborators: St. Olavs Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: OPI-14-001; 2014-001465-27 (EudraCT Number)
Record Dates: First submitted 2014-11-23; First posted 2014-12-04 (Estimated); Last update posted 2018-10-17 (Actual); Status verified 2018-10

CONDITIONS: Drug Overdose
Keywords: Emergency Treatment; Morphine Derivates; Heroin; Antidotes; Administration, Intranasal; Pharmacology; Naloxone; Healthy volunteers
MeSH Terms: conditions — Drug Overdose | interventions — Remifentanil

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intranasal naloxone (Experimental): 8 mg/ml naloxone 0,1 mL IN as one puff in one nostril in supine position
  Interventions: Drug: Intranasal naloxone; Drug: Remifentanil; Device: Aptar Unidose
- Intramuscular naloxone (Active Comparator): 0,4 mg/ml Naloxone B Braun 2 ML in deltoid muscle
  Interventions: Drug: Intramuscular naloxone; Drug: Remifentanil

INTERVENTIONS:
Drug: Intranasal naloxone — Administer 0,1 ml 8 mg/ml naloxone intranasally, dose = 0,8 mg naloxone
  Arms: intranasal naloxone
Drug: Intramuscular naloxone — Administer 2 mL, dose intramuscular naloxone 0,8 mg
  Other Names: Naloxone B Braun 0,4 mg/ml
  Arms: Intramuscular naloxone
Drug: Remifentanil — Administer remifentanil intravenously by way of Target Control Infusion, Minto model at a target of 2,5 ng/ml. This to achieve a state of safe and predictable opioid influence to assess pharmacodynamic response to naloxone. After treatment of 4 participants protocol amended 22. january 2015 to reduce remifentanil target to 1,25 ng/ml in the next 4. In the last 4 participants the dose will be decided later, but not exceed 2,5 ng/ml.
Device: Aptar Unidose — This is the spray device chosen, and its function in this setting (spray up side down) will be assessed by weighing the device before and after administration.
  Arms: intranasal naloxone

SUMMARY:
Overdose with potential deadly outcome is a serious problem among opioid abusers, not least in Norway. The annual death toll from overdose is about 250, higher than road traffic accidents. Those who inject heroin or other opioids are considered to have the highest risk for death from overdose. To save lives, immediate treatment with a μ-opioid antidote such as naloxone is required. Usually naloxone is injected into a muscle or a blood vessel. Administration of naloxone via the nose (intranasal) has been suggested as an alternative for use by emergency teams and possibly also bystanders. This is not only an easier way to give naloxone, but would also eliminate the risk for needle stick injuries and blood contamination. In a series of studies on intranasal naloxone at The Norwegian University of Science and Technology, this study explores pharmacokinetics and pharmacodynamics of intranasal and intramuscular naloxone in healthy volunteers under the influence of remifentanil.

DETAILED DESCRIPTION:
Healthy volunteers will be brought into a state of opioid influence in a well-known, short acting, controlled and safe manner using remifentanil.

Naloxone is a well-known, well-tolerated drug with an excellent safety profile over many decades of use. The current formulation has proven safe and without local or systemic side effects in the studies conducted so far. The excipients in the present nasal formulation are all well known.

This study has two aims. Firstly to investigate what naloxone does to the body under opioid influence, applying a well-tested model with infusion of the potent opioid remifentanil (Target Control Infusion). This will create a state of strong opioid effect for a short time and in a highly controlled fashion, inducing a state of miosis, reduced respiratory rate and reduced sensation to pain, all three strong indicators of opiates. Naloxone will antagonise these effects, and this change can be measured. Choosing intramuscular 0.8 mg naloxone for comparison means that the novel intranasal naloxone formulation will be compared with the well-established and described treatment protocol for opioid overdose in Norway used today.

Secondly the pharmacokinetic profile of intranasal and intramuscular naloxone will be studied. The same measurements as in preparative studies (OPI 12-001 and OPI 13-001) will be taken: Serum naloxone concentration over time to calculate maximum concentration, Time to maximum concentration, Area Under the Curve and Relative bioavailability. There are two main reasons to repeat these measurements. In contrast to the previous studies under the current protocol the participants will be under the influence by strong opioids. This may have significant physiologic effects, and it will be explored whether the pharmacokinetics of the intranasal formulation are changed. The other reason is that in this study pharmacokinetics of naloxone will be compared with the actual dosage and administration routes of naloxone as used by doctors and paramedics in the pre-hospital setting. This has not been done before, in spite of the widespread use of this treatment, The measurements of remifentanil in serum open the possibility to relate pharmacodynamic data directly to an actual serum concentration of the opioid at the same time.

Care will be taken not to include opioid users in this study as naloxone would precipitate acute withdrawal. Also possible drug misusers will be excluded as well as people who have access to remifentanil and infusion equipment in their daily work, although the abuse potential of this highly specialised drug is minimal.

Safety of the formulation will also be studied by measuring vital signs and for the patient to report any nasal discomfort or potential adverse reactions during the study.

By weighing spray device, and intramuscular syringes before and after discharge the reliability of the dose delivered will be confirmed.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists (ASA) class I
* ECG without pathologic abnormalities
* BMI range of 18,5 - 24,9 kg/m2.
* lab values within reference values at St Olav's Hospital for the relevant haematological and biochemical test for inclusion:

  * Haemoglobin (male: 13.4-17.0 g/dL, female 11.7 - 15.3 g/dL)
  * Creatinine (male: 60-105 micromole/L, female 45 - 90 micromole/L)
  * Aspartate aminotransferases (ASAT) (male: 15-45 U/L, female: 15-35 U/L)
  * Alanine transaminase (ALAT) (male: 10-70 U/L, female: 10-45 U/L)
  * Gamma glutamyl transpeptidase (GT) (male: 10-80 U/L, female: 10-45 U/L)
  * For women in reproductive age: serum HCG (normal under 3 ye/L)
* Signed informed consent and expected cooperation of the subjects for the treatment

Exclusion Criteria:

* Taking any medications including herbal medicines the last week prior to treatment visits
* Current or history of drug and/or alcohol abuse (To assess problematic drug or alcohol use we use the CAGE AID screening tool)
* History of contact with police or authorities in relation to alcohol or drug offences
* History of prolonged use of opioid analgesics
* History of prior drug allergy
* Having any local nasal disease or nasal surgery for the last 2 months or recent cold for the last week
* Pregnant women (HCG over 3 ye/L at inclusion)
* Women in reproductive age not using high efficacy contraceptives (Oral contraceptives, Patch (Evra), Implants, Vaginal ring, Hormonal IUD, Copper intra-uterine device (IUD), Sterilization) throughout the study period until their last visit.
* Breastfeeding women
* Participants with access to remifentanil or other potent opioids in their daily workplace.
* Hypersensitivity to naloxone or remifentanil hydrochloride and/or to any of its excipients.
* Any reason why, in the opinion of the investigator, the patient should not participate.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2014-12 (Actual); Primary Completion 2015-04 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Pharmacodynamic profile of naloxone- Heat Pain Threshold | 120 minutes
  We will measure time to maximum reversal, and duration of reversal of opioid effect on heat pain threshold measured. Heat pain thresholds will be tested using a Somedic MSA Thermotest (Somedic AB, Hørby, Sweden). This apparatus can measure the relationship between the intensity of controlled thermal stimuli and the associated perception. The stimulus (1 degree Celsius per sec rise time) is applied to the intact skin by a hand-held thermode while monitoring the temperature. The thermode (area 25x 50 mm= 12,5 cm2) will be placed over the non-dominant thenar eminence. Once the sensation changes from warm to painful the subject stops the increase in temperature by pressing a button, and the thermode cools down. The heat pain threshold (HPT) is measured in degrees C, and we will calculate the average of three repeated single HPTs.
Pharmacodynamic profile of naloxone. Pupillometry | 120 minutes
  Using a Neuroptics VIP 200 Pupillometer (Neuroptics, Irvine, CA, USA) we will measure the size of the pupils as a pharmacodynamic measure. The treatment visits will be conducted in a quiet room, with moderate, stable ambient lighting. Using a luxometer we will ensure similar light conditions in each visit of each participant. We will ask the participant to focus on a distant point in the room. The pupillometer will be placed over the measured eye and its position adjusted until the eye was correctly aligned within the LCD screen of the pupillometer. The reading will be recorded in CRF and/ or local work sheet A measurement of the pupils should take less than 10 seconds, and the result is given in millimetre, with an accuracy of 0.1mm and the results recorded. It is a non-invasive and pain free measurement.

SECONDARY OUTCOMES:
Adverse Events | minimum 6 days
  will be reported from the start of the first session to the follow-up visit.
Quantitate serum concentrations of remifentanil at specified time points | 110 minutes
  Measure serum concentration of remifentanil by Gas Chromatography-Mass Spectrometry (GCMS) at 0,15,30,45, 60 and 90 minutes.
Suitability of spray device in prehospital setting | 100 minutes
  By weighting spray device before and after intranasal administration to asses function in the supine patient.
Pharmacokinetics: Area Under the Curve of IN and IM naloxone | 360 minutes
  Measurement of serum naloxone at times 2,5,10,15,20,25,30,35,45,60,90,120,240 and 360 minutes after naloxone administration
Pharmacokinetics: maximum concentration (Cmax) of IN and IM naloxone | 360 minutes
  Measurement of serum naloxone at times 2, 5, 10, 15, 20, 25, 30, 35, 45, 60, 90, 120, 240 and 360 minutes after naloxone administration
Pharmacokinetics: time to maximum concentration (Tmax) of IN and IM naloxone | 360 minutes
  Measurement of serum naloxone at times 2, 5, 10, 15, 20, 25, 30, 35, 45, 60, 90, 120, 240 and 360 minutes after naloxone administration

CONTACTS AND LOCATIONS:
Overall Officials: Toril A Nagelhus Hernes, phd prof, Study Director — Norwegian University of Science and Technology
Locations (1):
- Department of Circulation and Medical Imaging, Trondheim, Norway

REFERENCES:
- [Result] Skulberg AK, Tylleskar I, Nilsen T, Skarra S, Salvesen O, Sand T, Loftsson T, Dale O. Pharmacokinetics and -dynamics of intramuscular and intranasal naloxone: an explorative study in healthy volunteers. Eur J Clin Pharmacol. 2018 Jul;74(7):873-883. doi: 10.1007/s00228-018-2443-3. Epub 2018 Mar 22. PMID 29568976